CLINICAL TRIAL: NCT01682304
Title: Observational Study of Epigenomic Dysregulation in Preeclampsia-Associated Chronic Hypertension
Brief Title: Epigenomic Dysregulation in Preeclampsia-Associated Chronic Hypertension
Status: Completed | Type: Observational
Sponsor: Ohio State University (Other)
Responsible Party: Principal Investigator, Cindy Anderson, PhD, WHNP-BC, FAAN, Ohio State University
Other Study IDs: GFHNRC611
Record Dates: First submitted 2012-09-05; First posted 2012-09-10 (Estimated); Last update posted 2022-10-12 (Actual); Status verified 2022-10

CONDITIONS: Preeclampsia; Hypertension; Pregnancy Induced Hypertension
Keywords: preeclampsia; hypertension; blood pressure; pregnancy induced hypertension; chronic hypertension
MeSH Terms: conditions — Pre-Eclampsia; Hypertension; Hypertension, Pregnancy-Induced

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Sputum and peripheral blood will be collected for DNA extraction and epigenetic analyses.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- History of Preeclampsia: Chronic hypertension with history of preeclampsia Chronic hypertension without history of preeclampsia

SUMMARY:
Preliminary data from the investigator's lab identified novel patterns of differential DNA methylation in genes regulating cardiovascular and metabolic function in blood from women during the first trimester of pregnancy who were destined to develop preeclampsia (PE) in the third trimester. Further, common patterns of differential DNA methylation were found in the common genes from placental tissue at time of birth in the same women after diagnosis with PE, suggesting that the epigenomic patterns that predict pregnancy-induced hypertension may also underlie the development of chronic hypertension years after.

It is unknown whether aberrant DNA methylation in pregnancy-induced hypertension is the mechanism by which chronic hypertension develops in these women remote from pregnancy nor is it known if hypertension remote from PE is as responsive to therapeutic treatment of hypertension compared to women who develop hypertension without history of PE. The investigators plan to objectively test the central hypothesis and attain the objective of this project

DETAILED DESCRIPTION:
Women comprise 51% of the total heart disease deaths in the United States (NC with an estimated economic cost expected to climb to more than $258 billion. Hypertension, a prevalent manifestation of early cardiovascular disease, is a silent condition that contributes to significant adverse health consequences. Preeclampsia (PE), a form of pregnancy-induced hypertension diagnosed in the second half of pregnancy, is now established as a non-modifiable risk factor for future development of hypertension. As PE carries a familial risk for future development of PE in female offspring, the implications of increased risk for PE-associated future development of chronic hypertension further compounds the significance of this unique cardiovascular risk. This raises an important health concern, though little is known about the mechanisms underlying risk of PE-associated future chronic hypertension. As epigenetic patterns of DNA methylation are associated with transfer across generations and are known to be dysregulated in PE, we propose to test the central hypothesis that differential DNA methylation patterns in key cardiovascular genes identified in women with PE serve as a biomarker and predictor for therapeutic responsiveness for the remote diagnosis and prognosis of chronic hypertension, respectively. Therefore, the purpose of this study is to identify distinct epigenetic patterns of DNA methylation associated with preeclampsia (PE) that underlie the future development of hypertension and to determine the implication on responses to moderators and therapeutic interventions in the management of chronic hypertension.Univariate analysis of variance will be used to test associations between DNA methylation in genes and chronic hypertension among women with and without a history of preeclampsia. We will use multiple linear regression to examine differences in treatment responses to high blood pressure based on DNA methylation patterns in candidate cardiovascular genes.

ELIGIBILITY:
Inclusion Criteria:

* Female gender
* history of prior pregnancy
* diagnosis of chronic hypertension
* current treatment of chronic hypertension
* age 30 - 50 years old

Exclusion Criteria:

* presence of comorbid conditions that influence cardiovascular health (SLE, congenital cardiac anomalies

Ages: 30 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Females diagnosed with chronic hypertension with a prior pregnancy
Sampling Method: Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2012-05; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
DNA methylation pattern | age 30-65
  Determine DNA methylatiion patterns in women with hypertension who have/have not had a prior diagnosis of preeclampsia

SECONDARY OUTCOMES:
Vascular function | aged 30-65
  Determine differences in vascular function among women aged 30-65, diagnosed with hypertension and who have/have not had a prior diagnosis of preeclampsia

CONTACTS AND LOCATIONS:
Overall Officials: Cindy M Anderson, PhD, Principal Investigator — Ohio State University
Locations (1):
- The Ohio State University, Columbus, Ohio, United States